CLINICAL TRIAL: NCT02828241
Title: A Multi-center, Randomized, Double-Blind, Parallel-group, Placebo-Controlled Study to Assess the Efficacy, Safety and Tolerability of DFD-04 (Itraconazole) Ointment, 5% in Patients With Inflammatory Lesions of Rosacea Over 12 Weeks
Brief Title: A Study to Assess the Efficacy, Safety and Tolerability of DFD-04
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DFD04-CD-002
Record Dates: First submitted 2016-07-07; First posted 2016-07-11 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DFD-04 Ointment (Experimental): DFD-04 (Itraconazole) Ointment
  Interventions: Drug: DFD-04 Ointment
- Placebo Ointment (Placebo Comparator): Placebo Ointment
  Interventions: Other: Placebo Ointment

INTERVENTIONS:
Drug: DFD-04 Ointment
  Arms: DFD-04 Ointment
Other: Placebo Ointment
  Other Names: Placebo
  Arms: Placebo Ointment

SUMMARY:
The purpose of this exploratory study is to assess the efficacy, safety and tolerability of DFD-04 Ointment for topical treatment of rosacea over 12 weeks of treatment.

DETAILED DESCRIPTION:
Subjects with mild to moderate papulopustular rosacea (Investigator's Global Assessment [IGA] grade 2-3), a Clinician's Erythema Assessment (CEA) score of 2-3 and 6-30 inflammatory lesions (papules and pustules) were randomized to treatment with DFD-04 ointment or Vehicle ointment in a ratio of 2:1.

During the 12-week treatment period subjects used the IMP twice daily with approximately 12 hours between applications. Subjects were instructed to treat affected skin in a defined treatment area on the face.

The investigator assessed efficacy by using an IGA 5-point scale and CEA 4-point scale and by counting the number of inflammatory lesions on the face at Baseline (Day 1) and Weeks 4, 8 and 12 (End of Treatment [EoT], defined as complete clearance of inflammatory lesions or Week 12, whichever was earlier). Furthermore, a non-invasive biomarker assessment was done by using a Transdermal Analysis Patch (TAP) at Baseline (Day 1) and Weeks 4 and 12.

Safety assessments included investigator's assessment of application site reactions at Baseline (Day 1) and Weeks 4, 8, and 12 for all treated areas.

Other safety assessments included vital signs (blood pressure [BP] and pulse rate) and urine pregnancy tests (UPTs) (only for females), clinical laboratory parameters (serum and urine), extent of exposure, and Adverse Events.

In addition, pharmacokinetic (PK) analysis was performed to evaluate the systemic exposures of itraconazole and its active metabolite, hydroxyl-itraconazole, with blood samples drawn from the first 12 subjects at various pre-specified timepoints.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand the requirements of the study and be willing to give written informed consent.
2. Subjects must be willing to provide authorization to use protected health information.
3. Subjects, any gender or race, must be in good general health as determined by the Investigator
4. Subjects must have a clinical diagnosis of papulopustular rosacea, Investigator's Global Assessment (IGA) grade 2 - 3.
5. Subjects must have 6 - 30 inflammatory lesions (papules and pustules) of rosacea over the face.
6. Subjects must have a Clinician's Erythema Assessment (CEA) score of 2 - 3.
7. Subjects must have no more than 2 nodules.
8. Subjects must agree to only use the study products and to not use any other treatment for rosacea (prescription or over the counter) or any other skin care or cosmetics product (make-up etc.) on the facial skin of the treatment area during the course of the study.
9. Subjects must be free of any systemic or dermatologic disorder, which in the opinion of the Investigator, will interfere with the study results.
10. Females have a negative urine pregnancy test at the Screening and Baseline Visit.
11. Females must either be postmenopausal with no menses for at least 12 months or surgically sterile (hysterectomy or tubal ligation) or agree to use a reliable method of contraception with a failure rate of less than 1 percent per year when used consistently and correctly.
12. Subject must be in good general health as determined by the investigator and supported by the medical history and normal or not clinically significant abnormal vital signs (blood pressure and pulse).
13. Subject is physically able to apply study product to all affected areas.

Exclusion Criteria:

1. Females who are pregnant or nursing or planning to become pregnant during the study.
2. Subjects who have been treated for rosacea within the 30 days prior to the Baseline Visit.
3. Subjects who have been treated with systemic retinoids within 6 months prior to the Baseline visit.
4. Subjects who have participated in a trial involving any investigational product in the 30 days prior to the Baseline Visit.
5. Subjects with any disease or medical condition that would interfere with the study or place the subject at undue risk especially cardiovascular diseases, reduced lung function (including asthma), renal dysfunction or liver dysfunction.
6. Subjects who have been treated within 30 days prior to baseline visit with methadone,disopyramide, dofetilide, dronedarone, quinidine, ergot alkaloids (such as dihydroergotamine, ergometrine (ergonovine), ergotamine, methylergometrine (methylergonovine)), irinotecan, lurasidone, oral midazolam, pimozide, triazolam, felodipine, nisoldipine, ranolazine, eplerenone, cisapride, lovastatin, simvastatin, ticagrelor, terfenadine, astemizole, mizolastine, eletriptan, as well as lovastatin, simvastatin and atorvastatin and, in subjects with varying degrees of renal or hepatic impairment, colchicine, fesoterodine, telithromycin and solifenacin.
7. Subjects who use or have used systemic steroids within the 30 days prior to the Baseline Visit or any other immunosuppressive medication.
8. Subjects positive for human immunodeficiency virus (HIV), hepatitis B and hepatitis C-test at screening.
9. Subjects who are unable to comply with study requirements.
10. Subjects with other skin diseases that may confound the evaluation of rosacea.
11. History of organ transplant requiring immunosuppression, HIV, or other immune compromised state.
12. Subject who in the opinion of the investigator or physician performing the initial examination the subject should not participate in the trial, e.g. due to probable noncompliance or inability to understand the trial and give adequately informed consent
13. Subject with close affiliation with the investigator (e.g. a close relative) or persons working at the respective trial sites or subject who are an employee of sponsor.
14. Subject institutionalized because of legal or regulatory order.
15. History of drug or alcohol abuse in the last year.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas R Sidgiddi, MD, Study Director — Dr. Reddy's Laboratories Inc.
Locations (8):
- Germany (8):
  - Site 201, Berlin
  - Site 208, Berlin
  - Site 202, Bochum
  - Site 205, Hamburg
  - Site 203, Mahlow
  - Site 204, Münster
  - Site 207, Potsdam
  - Site 206, Wiesbaden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized to either DFD-04 Ointment or Placebo Ointment in a ratio of 2:1
Groups:
- DFD-04 Ointment: DFD-04 (Itraconazole) Ointment applied over the affected areas on the face twice daily with approximately 12 hours between applications.
- Placebo Ointment: Placebo Ointment applied over the affected areas on the face twice daily with approximately 12 hours between applications.
Period: Overall Study
Arm/Group | DFD-04 Ointment | Placebo Ointment
Started | 38 | 23
Completed | 30 | 21
Not Completed | 8 | 2
Not completed — Adverse Event | 7 | 2
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo Ointment: Placebo Ointment
  t
- Total: Total of all reporting groups
Arm/Group | DFD-04 Ointment | Placebo Ointment | Total
Number analyzed (Participants) | 38 | 23 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (8.1) | 44.3 (10.2) | 48.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 18 | 43
  Male | 13 | 5 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 23 | 61
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 38 | 23 | 61

OUTCOME MEASURES:

1. Primary Outcome: Change in Inflammatory Lesion Counts
Description: Mean change from Baseline in the inflammatory lesion count at the End of Treatment. A lower score at the end of the study compared to Baseline is considered a better outcome.
Time Frame: At the end of study (12 weeks)
Population: Intent to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Number of lesions
Arm/Group | DFD-04 Ointment | Placebo Ointment
Number analyzed (Participants) | 38 | 23
Number of lesions | -1.4 (13.8) | 2.9 (17.5)

2. Primary Outcome: Number of Subjects With Investigator's Global Assessment (IGA) Success
Description: Number of subjects with treatment success based on Investigator's Global Assessment (IGA) score at the End of Treatment, defined as an IGA score of 0 (clear) or 1 (almost clear) with composite grade change from Baseline of at least 2 points.
Time Frame: At the end of study (12 weeks)
Population: Intent to Treat (ITT) population
Measure: Number; unit: participants
Arm/Group | DFD-04 Ointment | Placebo Ointment
Number analyzed (Participants) | 38 | 23
participants | 3 | 2

3. Primary Outcome: Number of Subjects With Treatment Success by Clinician's Erythema Assessment (CEA) Scale
Description: Number of subjects with Treatment Success defined as a score of 0 or 1 and a 2 grade improvement on the CEA scale from Baseline to 12 weeks.
Time Frame: At end of study (12 weeks)
Population: ITT population
Measure: Number; unit: participants
Arm/Group | DFD-04 Ointment | Placebo Ointment
Number analyzed (Participants) | 38 | 23
participants | 2 | 2

ADVERSE EVENTS:
Time Frame: From start of treatment until the end of study visit at 12 weeks.
Arm/Group | DFD-04 Ointment | Placebo Ointment
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/23
Other Adverse Events (participants affected / at risk) | 37/38 | 19/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DFD-04 Ointment (N=38) | Placebo Ointment (N=23)
Any Gastrointestinal Disorder (Gastrointestinal disorders) | 4 (7) | 3 (6)
Any General Disorder and Administrative Site Condition (General disorders) | 29 (127) | 13 (36)
Any Infections and Infestations (Infections and infestations) | 12 (16) | 7 (11)
Any Investigations (Investigations) | 2 (5) | 1 (1)
Any Musculoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 6 (9) | 2 (2)
Any Skin and Subcutaneous Tissue Disorders (Skin and subcutaneous tissue disorders) | 7 (13) | 5 (6)
Toothache (Gastrointestinal disorders) | 2 (4) | 0 (0)
Application Site Dryness (General disorders) | 7 (7) | 2 (2)
Application Site Erythema (General disorders) | 10 (13) | 4 (4)
Application Site Exfoliation (General disorders) | 5 (5) | 4 (4)
Application Site Pain (General disorders) | 22 (46) | 7 (13)
Application Site Pruritus (General disorders) | 21 (42) | 9 (9)
Application Site Reaction (General disorders) | 6 (6) | 1 (1)
Application Site Pustules (Infections and infestations) | 2 (2) | 0 (0)
Bronchitis Bacterial (Infections and infestations) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (7) | 5 (6)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin Burning Sensation (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin Reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Phase 2 pilot study so sample size was small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No